CLINICAL TRIAL: NCT07341984
Title: Individualized Physiotherapy Addressing Patient-Specific Deficits in Amyotrophic Lateral Sclerosis Compared to Usual Care Physiotherapy: A Prospective, Pseudorandomized, Controlled, Interventional Study
Brief Title: A Physiotherapy Intervention Study in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: Train ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charlotte Vogt (Other)
Responsible Party: Sponsor-Investigator, Charlotte Vogt, Sponsor-Investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BASEC 2025-02230
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Physiotherapy Group (Experimental): This group receives an individualized physiotherapy program tailored to patient-specific functional deficits. Two thrids of participants are allocated to the intervention group.
  Interventions: Other: Individualized Physiotherapy
- Usual Care Physiotherapy Group (Active Comparator): This group continues to receive usual care physiotherapy in accordance with standard clinical practice. One third of participants are allocated to the control group.
  Interventions: Other: Individualized Physiotherapy

INTERVENTIONS:
Other: Individualized Physiotherapy — see above

SUMMARY:
This study investigates whether an individualized physiotherapy program, tailored to each patient's specific motor deficits, can better support physical function compared with usual care physiotherapy in people with ALS.

The individualized program is guided by diagnostic assessments using a robotic leg press system, which helps identify strengths and weaknesses in muscle function and movement control.

Participants will receive either individualized physiotherapy or standard physiotherapy and will be followed for 12 months. The aim of the study is to improve physiotherapy strategies for people with ALS in a safe and patient-centered manner.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of clinically probable, probable laboratory-supported, or definite ALS (revised El Escorial criteria) or upper motor neuron only (OPM classification [onset, propagation, motoneuron involvement])
* age ≥18 years; ability to understand study information and provide written informed consent
* Willingness and ability to perform individualized exercise according to the study protocol (approximately three to five sessions of 30 minutes per week) for the duration of the intervention period
* Individuals of all sexes and gender identities are eligible for inclusion

Exclusion Criteria:

* pregnancy, tracheostomy, continuous assisted ventilation, or other significant non-ALS pulmonary disease
* other neurodegenerative or neuromuscular conditions that may confound assessments
* concomitant life-threatening disease or impairment interfering with functional assessment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Climbing stairs (ALSFRS-R [amyotrophic lateral sclerosis functional rating scale - revised] - item 9: score range 0 to 4 with 4 indicating normal function) | 6 months
  funcitonal

CONTACTS AND LOCATIONS:
Locations (1):
- ALS Clinic, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No